CLINICAL TRIAL: NCT02960035
Title: A Prospective Study of the Use of the Madrid Ultrasound Scoring System in the Treatment of Anti-TNF Blocker to Peripheral Tendonitis in Patients With Spondyloarthritis
Brief Title: A Study of the MASEI in the Treatment of Anti-TNF Blocker to Peripheral Tendonitis in Patients With Spondyloarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Prof, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: [2015]2-158
Record Dates: First submitted 2016-10-06; First posted 2016-11-09 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Spondyloarthropathy
Keywords: Mardird sonographic enthesis index; Spondyloarthropathy; Ultrasonics; Etanercept
MeSH Terms: conditions — Spondylarthropathies | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- etanercept 50mg/week (Experimental): Patients who entered the study continued on the same NSAIDs medications. The NSAIDs dose was kept unchanged throughout the study. All patients were provided with the once-weekly 50 mg dose in the form of etanercept for 24 weeks. After 24 weeks, those patients who had maintained a ASDAS-CRP ≤2.1 during period 1 will be randomised to one of three arms (period 2): this arms will receive ETN 50 mg weekly (unchanged). In all three arms, the patients continued NSAIDs, and other medications, at the same dose.
  Interventions: Drug: 50mg etanercept
- etanercept 25mg/week (Experimental): Patients who entered the study continued on the same NSAIDs medications. The NSAIDs dose was kept unchanged throughout the study. All patients were provided with the once-weekly 50 mg dose in the form of etanercept for 24 weeks. After 24 weeks, those patients who had maintained a ASDAS-CRP ≤2.1 during period 1 were randomised to one of three arms (period 2): this arms will receive ETN 25 mg weekly (half dose). In all three arms, the patients continued NSAIDs, and other medications, at the same dose.
  Interventions: Drug: 25mg etanercept
- PLACEBO (Placebo Comparator): Patients who entered the study continued on the same NSAIDs medications. The NSAIDs dose was kept unchanged throughout the study. All patients were provided with the once-weekly 50 mg dose in the form of etanercept for 24 weeks. After 24 weeks, those patients who had maintained a ASDAS-CRP ≤2.1 during period 1 were randomised to one of three arms (period 2): this arms will receive placebo weekly. In all three arms, the patients continued NSAIDs, and other medications, at the same dose.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 50mg etanercept — Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injection, 50mg per week
  Other Names: 50mg Yisaipu®
  Arms: etanercept 50mg/week
Drug: 25mg etanercept — Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc Fusion Protein Injection, 25mg per week
  Other Names: 25mg Yisaipu®
  Arms: etanercept 25mg/week
Drug: placebo
  Arms: PLACEBO

SUMMARY:
This is a randomized, double-blind, multicentral clinical trial to investigate the efficacy of Recombinant Human Tumor Necrosis Factor-α Receptor Ⅱ IgG Fc fusion protein injection (Yisaipu®) in the treatment of peripheral enthesitis in active axial spondyloarthritis(SpA) patients.

DETAILED DESCRIPTION:
Mardird sonographic enthesis index (MASEI) was one of the most wide used scoring systems for peripheral enthesitis and the only one based on OMERACT definition of enthesopathy by EULAR. The primary purpose is to assess the MASEI to discover the value of US in diagnosis and prognosis. The second prupose is to assess different maintaining treatment programme in SpA patients with improvement of MASEI. The trial will include 96 patients with stable NSAIDs therapy, and at the first stage they will receive 24-week full-dose of Yisaipu®. Then at the second stage the patients who achieve low disease activity (LDA, ASDAS<2.1) at 24th week will be randomizedly divided into three group: full-dose of Yisaipu® group, half-dose of Yisaipu® group and placebo group. And the blind stage will last for 24 weeks. Patients who complete the 48-week therapy or achieve disease-flare criteria during the blind stage would finish the study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the 2009 ASAS criteria for axial spondyloarthritis(SpA), and without bilateral more than grave 2 or unilateral more than grave 3 sacroilitis on X ray plan
* Active disease phase of SpA, defined as BASDAI≥4 or ASDAS≥2.1
* Inadequate response to NSAID≥4 week
* Application of NSAID with stable dose for no less than 2 weeks
* Stable dose of prenisone for at least four weeks at ≤10mg per day if used at screening, or stop use for at least 4 weeks
* Stable dose of any DMARD for at least four weeks if used at screening, or stop use for at least 4 weeks
* Stop and receiving washing out for at least 4 week if receiving Chinese traditional drug for AS, physical treatment, vaccication or IVIG
* The lab exam should achieve the criteria as below:

  * Hb ≥ 85g/L
  * 3.5×109/L ≤ WBC count ≤ 10×109/L
  * PLT ≥ lower limit of normal range
  * ALT ≤ 2 fold of upper limit of normal range
  * serum creatine ≤ upper limit of normal range
* Negative pregnacy test for female patients. And promise to carry out contraception during the trial and 6 weeks after the trial is ended
* Sign the informed consent

Exclusion Criteria:

* Previous application of any biologic agents
* Allergic to any element of Yisaipu®
* Intolerance to NASID
* History of active tubercolosis, or radiographic evidence of present or previous history of pulmonary tubercolosis, or close contact with patients with tubercolosis, or with high risk of infection of tubercolosis such as immune suppression status, or strong positive of PPD skin test with diameter ≥10mm
* Presence of acute infection or acute onset of chronic infection at screen
* Invasive fungal infection or conditional infection within 6 months prior to screen
* Present or history of serious liver disease
* History of infection on artifitial joints
* Organ transplantation surgery within 6 months prior to screen
* Presence of other autoimmune diseases, including IBD, psoriasis, uveitis, SLE, multiple sclerosis, etc
* History of congestive heart failure
* History of malignancies within 5 years prior to screen, excluding complete resection of squamous cell carcinoma, or basal cell carcinoma or cervical carcinoma in situ
* AIDS or HIV infection
* History of lymphoma or lymphoproliferative disorders
* Presence of serious disorder of important organs or system
* Presence of factors which may influence the compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The change of Mardird sonographic enthesis index (MASEI) at 24 weeks | 24 weeks
  The change of Mardird sonographic enthesis index (MASEI) from week 0 to week24

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Prof., Study Director — Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China